CLINICAL TRIAL: NCT05315518
Title: Effect of Using Shade Blocker Versus Chameleon Effect on Shade Matching of Two Single-shade Resin Composite Materials in Class IV Restorations: A One Year Randomized Clinical Trial
Brief Title: Effect of Using Shade Blocker Versus Chameleon Effect of Two Single Shade of Resin Composite in Class IV Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sarah ali mohamed ahmed, Master's degree student-faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPR 14/3/2022
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Discoloration, Tooth
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single shade universal resin composite (omnichroma) with blocker (Experimental): (OMNICHROMA BLOCKER) is indicated for preventing shade-matching interference in Class IV restorations, Masking dark dentition and dentin. In cases where there is a lack of tooth structure to bond to, (BLOCKER) works as a supplementary product to provide a lingual wall to the restoration, prevent shade-match obstruction and mask staining.
  Interventions: Diagnostic Test: single-shade universal resin composite (omnichroma) with blocker( omnichroma blocker)
- single shade universal resin composite(GC solare sculpt) with chameleon effect (Active Comparator): One-shade universal resin composite (GC solare sculpt) gives very natural appearance, High gloss retention over time, time saving regarding to layering technique, wide shade matching range (chameleon effect) and delivering lifelike aesthetic restorations. These features can be offered by supra-nano spherical filler which have controlled refractive index, records excellent esthetic properties in small and medium class IV restorations.
  Interventions: Diagnostic Test: single-shade universal resin composite (omnichroma) with blocker( omnichroma blocker)

INTERVENTIONS:
Diagnostic Test: single-shade universal resin composite (omnichroma) with blocker( omnichroma blocker) — (OMNICHROMA BLOCKER) is indicated for preventing shade-matching interference in Class IV restorations, Masking dark dentition and dentin. In cases where there is a lack of tooth structure to bond to, (BLOCKER) works as a supplementary product to provide a lingual wall to the restoration, prevent shade-match obstruction and mask staining.

SUMMARY:
Aim of this study will be conducted to compare the shade matching and clinical performance of shade blocker versus chameleon effect of two single-shade of universal resin composite in class IV restorations over 1 year evaluation period

DETAILED DESCRIPTION:
The color matching of both groups will be evaluated visually using modified USPH criteria

ELIGIBILITY:
Inclusion Criteria:

moderate class IV defect with no lingual wall presence of favorable occlusion and teeth are in normal contact with the adjacent teeth good oral hygiene cooperative patients

-

Exclusion Criteria:

* tooth hypersensitivity severe periodontal affection non vital teeth heavy smoking

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-09-05 (Estimated); Primary Completion 2022-10-05 (Estimated); Study Completion 2023-04-07 (Estimated)

PRIMARY OUTCOMES:
shade matching | 12 months
  the shade matching of both groups will be assessed visually by using modified USPH criteria.
  score: 1- Alpha : the restoration match the shade and translucency of the adjacent tooth 2-Bravo : there is a mismatch in the shade and translucency but it is within a normal range of tooth shade 3- Charlie: the mismatch is beyond the normal range of the tooth shade and translucency

CONTACTS AND LOCATIONS:
Overall Officials: sarah ahmed, master, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
The aim of the study is to compare the shade matching and clinical performance of shade blocker versus chameleon effect of two single-shade universal resin composite in class IV restorations over 1year evaluation period.
Supporting Information: Study Protocol
Time Frame: The restorations will be evaluated at T1= after 1 week T2= 3months T3= 6 months T4= 12 months
Access Criteria: * Patients with class IV defects (due to caries lesions, trauma…etc.)
  * Young adult (20 : 40 years old)
  * Good oral hygiene
  * Co-operative patients approving to participate in the study